CLINICAL TRIAL: NCT04727476
Title: The Use of Lisdexamfetamine in Clinical Practice at a Danish Child Psychiatric Outpatient Clinic Aimed at School Children (Age 7-13 Years) With Attention Deficit Disorders
Brief Title: The Use of Lisdexamfetamine for Children Aged 7-13 With Attention Deficit Disorders
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Nanna Roed Søndergaard, MD, Aarhus University Hospital
Other Study IDs: LDX-2013-2019; IIR-DNK-002529 (Other Grant/Funding Number: Takeda Pharma)
Record Dates: First submitted 2021-01-12; First posted 2021-01-27 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Attention Deficit Disorder; Attention Deficit Hyperactivity Disorder; Hyperkinetic Disorder
Keywords: ADHD; ADD; Lisdexamfetamine
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with attention deficit disorders: children aged 7-13 years who have attended a specialised outpatient clinic treating children with attention deficit disorders i in the period from 1 April 2013 to 5 November 2019.
  Interventions: Drug: Lisdexamfetamine

INTERVENTIONS:
Drug: Lisdexamfetamine — Prescription of lisdexamfetamine sometime during til period from 1 April 2013 to 5 November 2019.

SUMMARY:
Aiming at improving clinical practice regarding the use of lisdexamfetamine for the treatment of ADHD in children, the investigators want to retrospectively map the clinical use of lisdexamfetamine at a specialised outpatient clinic located at Aarhus University Hospital, Denmark treating children aged 7-13 with Attention Deficit Disorders in the period from 2013 to 2019. The investigators will describe the changes in prescription practice in the period, reported side effects and reasons for selecting and discontinuing treatment with lisdexamfetamine.

DETAILED DESCRIPTION:
Background

Attention deficit hyperactivity disorder (ADHD) is characterised by the core symptoms of inattention, hyperactivity and impulsivity, which are excessive for the person's age and developmental status. It is a clinical diagnosis based on observed and reported behavioural symptoms. Two main diagnostic systems are used currently, the International Classification of Diseases 10th revision (ICD-10) and the Diagnostic and Statistical Manual of Mental Disorders 5th edition (DSM-5). Both systems require presence of symptoms in several settings such as school, home life and leisure activities as well as the presence of functional impairment due to symptoms of ADHD (e.g. impairment of psychological, social and/or educational functioning). Symptoms should be evident in early life; for ICD-10 by age 7 and for DSM-5 by age 12. Overall, the diagnostic criteria of ADHD are less stringent according to DSM-5 compared to ICD-10, which is reflected by a higher prevalence of ADHD in populations where the DSM-5 diagnostic criteria are applied. A systematic review (Sayal et al.) from 2018 of 55 studies (25 from the USA, seven from the UK, and 23 outside the USA and UK) reported a prevalence of ADHD in children and adolescents varying from approximately two to seven percent depending mostly on the diagnostic criteria, making it one of the most common psychiatric disorders in children and adolescents.

In Denmark the ICD-10 diagnostic system is used. The National Institute for Health and Care Excellence (NICE) as well as The National Clinical Guidelines from the Danish Health Authority recommend pharmacological treatment for children and adolescents with moderate to severe ADHD. Severity is determined by a clinical assessment based on number of symptoms and functional impairment. Both guidelines recommend the use of methylphenidate (MPH) as the first choice of treatment. In the event that the use of MPH is non-effective in an adequate dosage or results in adverse effects, it is recommended to switch to atomoxetine (ATX), dexamfetamine (DX) or lisdexamfetamine (LDX). The subsequent choice of medication should take into consideration the adverse effect profiles and duration of effect of the different drugs as well as the reason for the switch.

In February 2013, Elvanse (LDX) received marketing authorization in the UK and Europe. It became available for sale for the treatment of ADHD in children and adolescents in Denmark in April 2013.

LDX is an inactive prodrug which is gradually activated to DX by means of peptidase enzymes in the red blood cells. Thus, LDX is a controlled-release drug where a single dose has an effect on the ADHD core symptoms for up to 13 hours. The formulation as a prodrug reduces its potential for abuse. According to www.medstat.dk which is based on data from the Danish Register of Medicinal Product Statistics (LSR), the sales of lisdexamfetamine has been steadily increasing during the years it has been on the market in Denmark.

In our clinical experience medical treatment of ADHD in children is often complicated by intolerable adverse effects (e.g. weight loss due to loss of appetite or disturbance of sleep), worsening of symptoms of comorbidities (e.g. anxiety, tic disorders or psychosis), lack of/inadequate effect or non-optimal day coverage of treatment. In our experience, these complications often lead to frequent switches in medical treatment. This is supported by a study by Ben Amor et al. (2014) in which the authors reported a one-year period prevalence of switching from one stimulant to either another stimulant, ATX or atypical antipsychotic of 19.5% in children and 17.4% in adolescents.

Another study by Warrer et al. (2016) reported that the mean duration of MPH treatment before switching to ATX was 11.2 months in a population of 55 children and adolescents aged 7-18 years with attention deficit disorders. 36% of the patients switched within the first 6 months, 56% within the first year and 76% within 1.5 years. 24% continued with MPH for 2.5 years before switching to ATX. The most common reasons for switching were adverse effects (78%), need for stable 24-hr effect (24%) or lack of effect (16%). The conclusion of this study as well as the conclusion of another study by Powell et al. (2011), was that the importance of continuously evaluating the treatment of the individual patient throughout the entire course of treatment needs to be emphasised, especially if there is no immediate good effect and tolerability of the first choice of medication.

Aiming at improving clinical practice regarding LDX, the investigators want to describe the changes in prescription practice in the period 2013 to 2019, reported side effects and reasons for selecting or discontinuing LDX. The investigators expect LDX to be prescribed more often in later years compared to earlier years because clinicians may be inclined to a select medical treatment they have experience with rather than a new one.

Hypotheses Hypothesis 1: The investigators expect LDX to be second choice in line with ATX in later years.

Hypothesis 2: The investigators expect the main reasons for switching to LDX to be adverse effects from MPH and/or ATX. The investigators expect to be able to describe top 5 adverse effects.

Hypothesis 3: The investigators expect patients who continue treatment with LDX to be comparable with patients who discontinue treatment with LDX regarding gender, age, diagnosis, ADHD symptoms at baseline and comorbidities.

Hypothesis 4: The investigators expect adverse effects to be the main reason for discontinuing LDX.

To our knowledge, there are no previous studies investigating the practical clinical use of LDX in Denmark.

Method

The study is a retrospective descriptive study that includes data from medical records of approximately 600 patients.

Patients will be identified in the electronic patient record system based on the inclusion criteria. Baseline data and outcome data will be extracted from medical records by Nanna Roed Søndergaard, MD, who will enter the data into a REDCap database designed for this purpose.

Patients will be categorised into three groups according to whether they have received treatment with LDX as a first, second or third choice of treatment. Combination treatment will also be registered.

Descriptive statistics will be used to summarise overall patient and treatment characteristics, duration of therapy to switches, clinical reasons for switches in therapy, clinical effect and adverse effects observed. Comparison between groups will be performed using parametric or non-parametric test. An alfa level will be set at 0.5 in all analyses. Analyses will be conducted using the statistical software program Stata 15.

In accordance with Danish legislation the study has been approved by the Danish Health and Medicines Authority, registered at the Danish Data Protection Agency and will be conducted in accordance with the Danish Act on Processing of Personal Data. This study requires no patient contact. It will not be possible to trace the results of the study back to individual patients. Data will be stored in MidtX in agreement with the EU General Data Protection Regulation (GDPR). According to Danish legislation, no ethics or institutional review board approvals are required for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 7-13 years at referral to the outpatient clinic.
2. Have been diagnosed with one or more of the following ICD-10 diagnoses: F90.0 Disturbance of activity and attention; F90.1 Hyperkinetic conduct disorder; F90.8 Other hyperkinetic disorders; F90.9 Hyperkinetic disorder, unspecified; F98.8 Other specified behavioural and emotional disorders with onset usually occurring in childhood and adolescence (attention deficit disorder without hyperactivity, excessive masturbation, nail-biting, nose-picking, thumb-sucking), F98.8C Attention deficit disorder without hyperactivity.

   Manual review of patients with the diagnosis F98.8 is deemed necessary to identify all patients with attention deficit disorder without hyperactivity due to changed diagnostic practice.
3. Prescription of lisdexamfetamine sometime during the period from 1 April 2013 to 5 November 2019.

Exclusion Criteria:

1. Prescribtion of ADHD medication prior to 1 April 2013.
2. Patients with the diagnosis F98.8 with the following denominations will be excluded; excessive masturbation, nail-biting, nose-picking, thumb-sucking.

Ages: 7 Years to 13 Years | Sex: All
Age Groups: Child
Study Population: The patients included in this study have attended a specialised outpatient clinic at the Department of Child and Adolescent Psychiatry at Aarhus University Hospital located in the Central Denmark Region. The specialised outpatient clinis treats children aged 7-13 years with moderate to severe ADHD. The catchment area of the Central Denmark Region comprises 1.3 million inhabitants. Patients are referred to the outpatient clinic from municipality services, general practitioners and to a lesser extent from other hospital units. The outpatient clinic is responsible for diagnosing and treating patients with the referral diagnosis of attention deficit disorder and comorbid conditions.
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Lisdexamfetamine as first, second and third choice of treatment (+/- dexamfetamine as supplementary treatment). | Prescription of lisdexamfetamine sometime during the period from 1 April 2013 until 5 November 2019.
  Number of patients receiving lisdexamfetamine as first, second and third choice (+/- dexamfetamine as supplementary treatment).

SECONDARY OUTCOMES:
Duration of treatment. | ADHD treatment prescribed in the period from 1 April 2013 to 5 November 2019.
  Duration of treatment of first, second and third choice of treatment (days/months).
ADHD symptoms. | At baseline and at the most stable dosage of a drug from prescription to discontinuation (first, second and third choice of treatment) in the period from 1 April to 5 November 2019..
  ADHD symptoms according to DuPaul's ADHD rating scale. The rating scale is sent out to parents and schools before each consultation every 6 months.
Adverse effects. | All adverse effects registered during medical treatment from prescription to discontinuation of a drug (first, second and third choice of treatment) in the period from 1 April 2013 to 5 November 2019.to .
  Adverse effects of the medical treatments registered by clinicians in the patient journals. Adverse effects will be classified by System Organ Class (SOC) and Preferred Term (PT) level according to the Medical Dictionary for Regulatory Activities (MedDRA) (International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use 2014.
Reasons for discontinuing medical treatment. | At the time point (date) when a medical treatment is discontinued in the period from 1 April 2013 to 5 November 2019..
  Reasons for discontinuing medical treatment (first, second and third choice of treatment) as registered by clinicians in the patient journals. Reasons will be categorised as being due to one or more of the following; lack of effect, adverse effects, patient/parental request, non-compliance, wish for more optimal day coverage.
Maximal dosage. | The maximal dosage prescribed of a drug from first prescription to discontinuation (first, second and third choice of treatment) in the period from 1 April to 5 November 2019.
  The maximal dosage of the prescribed drug from prescription to discontinuation of a medical treatment (first, second and third choice of treatment).
Final dosage. | Either the dosage immediately before switching medication or at the end of the study period (5 November 2019).
  Final dosage of a treatment.
Characteristics of patients continuing with lisdexamfetamine treatment. | In the period from 1 April 2013 to 5 November 2019
  Characteristics of patient continuing treatment with lisdexamfetamine regarding gender, age, diagnosis, ADHD symptoms at baseline, comorbidities, and adverse effect profile.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Roed Soendergaard, MD, Principal Investigator — Department of Child and Adolescent Psychiatry, Aarhus University Hospital, Denmark
Locations (1):
- Department of Child and Adolescent Psychiatry, Aarhus University Hospital, Aarhus, Region Midt, Denmark

IPD SHARING:
Plan to Share IPD: No